CLINICAL TRIAL: NCT05330481
Title: Exploring the Role of Body Mass in Exogenous Carbohydrate Oxidation Rates During Exercise
Brief Title: Body Weight and Carb Metabolism
Status: Completed | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Reader (Associate Professor) in Human Physiology, University of Bath
Other Study IDs: 6632
Record Dates: First submitted 2022-03-02; First posted 2022-04-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Exercise Metabolism
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- <70 kg body mass: Cyclists or triathletes with a body mass of less than 70 kg
  Interventions: Other: Moderate-intensity (relative) exercise with glucose ingestion
- >70 kg body mass: Cyclists or triathletes with a body mass of less than 70 kg
  Interventions: Other: Moderate-intensity (relative) exercise with glucose ingestion; Other: Moderate-intensity (absolute) exercise with glucose ingestion

INTERVENTIONS:
Other: Moderate-intensity (relative) exercise with glucose ingestion — 120 minutes of cycling at 95% of lactate threshold ingesting 90 g/h of glucose
Other: Moderate-intensity (absolute) exercise with glucose ingestion — 120 minutes of cycling at a power matched to participant in the <70 kg body mass group, ingesting 90 g/h of glucose
  Groups: >70 kg body mass

SUMMARY:
Whilst theoretically, body size should influence the capacity for intestinal carbohydrate absorption and thus exogenous oxidation rates during exercise, there is currently little empirical evidence to support this hypothesis. Accordingly, current nutrition guidelines for carbohydrate intake during exercise do not take body mass into account. Therefore, there is a need to establish whether body mass is related to exogenous carbohydrate oxidation rates during exercise. If such a relationship is established, this would lay the foundation to revise the current sports nutrition guidelines regarding carbohydrate intake during exercise.

The aims of this study are, therefore, to: 1) establish whether larger individuals display higher rates of exogenous carbohydrate oxidation than smaller individuals; and 2) establish if such a difference can be explained by the higher absolute exercise intensity, and thus the energy demand of exercise. It is hypothesised that larger individuals will demonstrate higher exogenous carbohydrate oxidation rates than smaller individuals, and that this difference will be partly (but not completely) diminished when the absolute intensity of exercise is matched.

ELIGIBILITY:
Inclusion Criteria:

* Able to cycle continuously for 2 hours at a moderate intensity
* VO2max of between 40-75 mL/kg/min
* Fat-mass index (determined by dual energy x-ray absorptiometry) < 5.5 kg·m-2

Exclusion Criteria:

* Diagnosed disorders of the gastrointestinal tract (e.g. crohn's, colitis etc.)
* People following a low-carbohydrate, high-fat diet
* Pregnant or lactating
* Diagnosed cardiovascular disease
* Possible symptoms of cardiovascular disease
* Diagnosis of diabetes of any type
* Hypercholesterolaemia (total cholesterol ≥ 6.2 mmol/L
* Hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
* Current smoker
* Family history of coronary artery disease (first-degree relative <60 years)
* Prevalence of vascular disease
* Autonomic neuropathy
* Kidney disease
* Diagnosed pulmonary disease (e.g. chronic obstructive pulmonary disease, asthma, interstitial lung disease or cystic fibrosis)
* Blood borne disease or infection
* Osteoporosis
* Osteoarthritis
* Blood clotting disorders
* Food intolerances/allergies (these may not specifically exclude you- please talk to the investigator)
* Sensitivity or allergy to anaesthetic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Trained cyclists or triathletes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Peak exogenous carbohydrate oxidation rate (g/min) | 120 minute
  Peak exogenous carbohydrate oxidation rate (g/min)
Total exogenous carbohydrate oxidation (g) | minutes 30-120 of exercise
  Sum of exogenous carbohydrate oxidation in g

SECONDARY OUTCOMES:
Total exogenous carbohydrate oxidation (g/kgFFM) | minutes 30-120 of exercise i
  Sum of exogenous carbohydrate oxidation (g/kgFFM)
Whole-body carbohydrate oxidation rate (g) | minutes 30-120 of exercise
  Sum of whole-body carbohydrate oxidation (g)
Whole-body carbohydrate oxidation rate (mg/kgFFM) | Sum of minutes 30-120 of exercise
  Sum of whole-body carbohydrate oxidation (mg/kgFFM)
Endogenous carbohydrate oxidation rate (g) | minutes 30-120 of exercise
  Sum of endogenous carbohydrate oxidation (g)
Endogenous carbohydrate oxidation rate (mg/kgFFM) | minutes 30-120 of exercise
  Sum of endogenous carbohydrate oxidation (mg/kgFFM)
Whole-body fat oxidation rate (g) | minutes 30-120 of exercise
  Sum of whole-body fat oxidation (g)
Whole-body fat oxidation rate (mg/kgFFM) | minutes 30-120 of exercise
  Sum of whole-body fat oxidation (mg/kgFFM)
Plasma lactate concentrations (mmol/L) | minutes 0-120 of exercise
  Plasma lactate concentrations (mmol/L)
Plasma glucose concentrations (mmol/L) | minutes 0-120 of exercise
  Plasma glucose concentrations (mmol/L)
Plasma non-esterified fatty acid concentrations (mmol/L) | minutes 0-120 of exercise
  Plasma non-esterified fatty acid concentrations (mmol/L)
Plasma insulin concentrations (pmol/L) | minutes 0-120 of exercise
  Plasma insulin concentrations (pmol/L)
Dietary carbohydrate intake (grams/day) | 72-hour food diary in g/d
  Dietary carbohydrate intake (grams/day)
Dietary sugar intake (grams/day) | 72-hour food diary
  Dietary sugar intake (grams/day)
Dietary fibre intake (grams/day) | 72-hour food diary
  Dietary fibre intake (grams/day)
Dietary fat intake (grams/day) | 72-hour food diary
  Dietary fat intake (grams/day)
Dietary protein intake (grams/day) | 72-hour food diary
  Dietary protein intake (grams/day)
Dietary energy intake (kiloJoules/day) | 72-hour food diary
  Dietary energy intake (kiloJoules/day)
Dietary energy intake (kilojoules/kilogram/day) | 72-hour food diary
  Dietary energy intake (kilojoules/kilogram/day)
Dietary carbohydrate intake (grams/kilogram/day) | 72-hour food diary
  Dietary carbohydrate intake (grams/kilogram/day)
Dietary sugar intake (grams/kilogram/day) | 72-hour food diary
  Dietary sugar intake (grams/kilogram/day)
Dietary fibre intake (grams/kilogram/day) | 72-hour food diary
  Dietary fibre intake (grams/kilogram/day)
Dietary fat intake (grams/kilogram/day) | 72-hour food diary
  Dietary fat intake (grams/kilogram/day)
Dietary protein intake (grams/kilogram/day) | 72-hour food diary
  Dietary protein intake (grams/kilogram/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom